CLINICAL TRIAL: NCT00299559
Title: An Open Clinical Cross-Over Trial to Compare the Kinetics of Etheric Oils Applied Onto the Skin or Via Smart Textiles
Brief Title: Kinetics of Etheric Oils, Smart Textiles vs. Ointment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EK222122005
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2007-11

CONDITIONS: Common Cold
Keywords: common cold; organic chemicals; menthol; cineole; camphor; etheric oils; alternative medicine; smart textiles
MeSH Terms: conditions — Common Cold | interventions — Camphor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): cross over application of both specimen
  Interventions: Drug: smart textiles containing menthol, camphor, cineol

INTERVENTIONS:
Drug: smart textiles containing menthol, camphor, cineol — application to skin

SUMMARY:
The purpose of the study is to determine whether the application form of etheric oils (camphor, cineol and menthol) causes changes in the concentration of this agents in the exhaled air. The second aim of the study is to determine differences in the subjective convenience of the application forms. We will test an commercial ointment application vs. smart textiles. Smart textiles are new high-tech products with the unique possibility to combine the textiles with functional products e.g. pharmaceutical agents.

DETAILED DESCRIPTION:
On the first appointment recruitment investigations will take place. After the person is enrolled to the study, the first determination of substances concentration in exhaled air and the convenience grade of the application form being exposed to will be achieved (study day 1). After a 7 days lasting washout phase on study day 2 newly determination of substances concentration and convenience grade of the other application will be assessed. Each study day will have an approximate duration of 11 h. During this time 9 samples of the persons exhaled air will be collected.

ELIGIBILITY:
Inclusion Criteria:

* caucasian
* Broca-index: between -20 and +25%
* who are willing and capable to confirm written consent to enrolment after ample information has been provided
* who are in a stable condition that it can be expected that no changes in relevant medical conditions will occur during the study.

Exclusion Criteria:

* subjects with any major relevant clinical abnormality (as based on extensive medical history, physical examination, vital signs)
* subjects with any major clinically relevant laboratory abnormality.
* subjects who participated in another trial with any investigational substance within the last 4 weeks
* subjects who smoke more than 15 cigarettes per day
* subjects who are known or suspected to be (social) drug dependent, incl. those drinking more than moderately and who are not willing to abstain from alcohol during the active study phase
* subjects who adhere to a diet or lifestyle (incl. competitive sports and weight lifting) that might interfere with the investigation
* subjects who are known or suspected not to comply with the study directives and/or who are known or suspected not to be reliable or trustworthy
* subjects who are known or suspected not to be capable of understanding and evaluating the information that is given to them as part of the formal information policy (informed consent), in particular regarding the risks and discomfort to which they would agree to be exposed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-03; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Determination of agents concentration in exhaled air on study day 1+2. On each day 9 samples of exhaled air will be obtained. | 24 h

SECONDARY OUTCOMES:
Grade of convenience of each application form will obtained at the end of each study day | 48 h

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Siegert, MDDPharm,PhD, Principal Investigator — Department of clinical Pharmacology, Medical Faculty Carl Gustav Carus, University of Technology
Locations (1):
- Department of clinical Pharmacology, Medical faculty Carl Gustav Carus, University of Technology Dresden, Dresden, Germany